CLINICAL TRIAL: NCT05707936
Title: Normal Saline Versus Heparin Intermittent Flushing for the Prevention of Occlusion in Port-a-Cath: Randomized Controlled Trial
Brief Title: Normal Saline Versus Heparin Intermittent Flushing for the Prevention of Occlusion in Port-a-Cath
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: CMRPVVM0141
Record Dates: First submitted 2022-10-28; First posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2022-10

CONDITIONS: Port-a-cath Occlusion; Normal Saline; Heparin Lock

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normal saline 20 ml (Experimental)
  Interventions: Drug: Normal Saline Flush 20 ml
- Normal saline 10 ml (Experimental)
  Interventions: Drug: Normal Saline Flush 10 ml
- usual care (heparin) (Active Comparator)
  Interventions: Drug: Heparin Flush (1000 USP, 10ml)

INTERVENTIONS:
Drug: Normal Saline Flush 20 ml — Normal Saline Flush 20 ml
  Arms: Normal saline 20 ml
Drug: Normal Saline Flush 10 ml — Normal Saline Flush 10 ml
  Arms: Normal saline 10 ml
Drug: Heparin Flush (1000 USP, 10ml) — Heparin Flush (1000 USP, 10ml)
  Arms: usual care (heparin)

SUMMARY:
Purpose:

An evidence implementation of a randomized controlled trial for whether there is the difference in intermittent flushing 0.9% normal saline and heparin? Design: a single-blind randomized controlled trial

Method:

This study is based on the 5A (Ask, Acquire, Appraise, Apply, Audit) of evidence health care step, and design randomized controlled trial for evidence implementation.

We will include inpatients over 20 years-old adults in New Taipei City TuCheng Hospital, Taiwan, who need administration medicine by port-a-catcher. The sample size is 192 according to G-power software. Random allocation software has using for block randomization, would assign to group A: flushing with 0.9% normal saline 10ml, group B: flushing with 0.9% normal saline 20ml, and group C: flushing with heparin 100 USP/ml. SPSS 20.0 software for statistical analysis, mean or standard deviation, one- way ANOVA would use.

ELIGIBILITY:
Inclusion Criteria:

Non-pediatric inpatients over 20 years of age with PAC placed for any disease and who need medication during hospitalization.

Exclusion Criteria:

History of PAC obstruction, continuous high volume drip via PAC, taking anticoagulant or antiplatelet agents, abnormal blood coagulation, pregnancy or contraceptive use, specified flushing solution by case

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
port-a-cath occlusion | in hospitalized (during admission), up to 12 weeks
  failure to infusion fluid
port-a-cath infection | in hospitalized (during admission), up to 12 weeks
  blood culture from port-A show bacterial growth